CLINICAL TRIAL: NCT04594746
Title: Oral Amiodarone for Acute Cardioversion of Atrial Fibrillation Study
Acronym: AAA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: we couldn't recruit enough participants
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB20-1555
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Amiodarone
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Drug and placebo will be encapsulated and blinded by the investigational pharmacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Amiodarone (Experimental): Amiodarone hydrochloride 2000 mg
  Interventions: Drug: Amiodarone Hydrochloride
- Placebo (Placebo Comparator): Oral placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amiodarone Hydrochloride — Amiodarone hydrochloride 2000 mg PO to be given as a 10-capsule dose pack and ingested in a single sitting with food
  Other Names: Cordarone; Nexterone
  Arms: Oral Amiodarone
Drug: Placebo — Oral placebo to be given as a 10-capsule dose pack and ingested in a single sitting with food
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The investigators will seek to determine the safety and efficacy of high-dose amiodarone (2000mg), given as a single uniform oral dose, for the treatment of acute atrial fibrillation in both a hospital inpatient and ambulatory outpatient setting. The investigators will conduct a placebo-controlled randomized trial, with outcome ascertainment at 48h.

DETAILED DESCRIPTION:
Background: Atrial fibrillation (AF) is estimated to affect over 33 million people worldwide and is often associated with significant co-morbidities such as myocardial infarction, heart failure, dementia, and embolic stroke. Consequently, AF poses a significant burden to the healthcare system, in both direct and indirect costs of disease.

The management of AF in the acute setting is complex, especially for patients who suffer from persistent AF, defined as sustained AF for > 7 days. While one possible treatment strategy involves allowing AF to continue whilst controlling the ventricular rate (i.e. rate control), in certain cases, it is preferable to terminate the AF and restore normal sinus rhythm (i.e. rhythm control) for relief of intolerable symptoms associated with AF.

There are several methods currently in use for rhythm control, including observation without intervention, use of oral and/or intravenous anti-arrhythmic drugs for pharmacological cardioversion, and electrical cardioversion. However, each of these strategies come with significant limitations. Amiodarone was originally developed for treatment of angina, but is now widely recognized for its anti-arrhythmic properties. Current American College of Cardiology/American Heart Association/European Society of Cardiology guidelines recommend the use of amiodarone as a cardioversion agent in both intravenous and oral administration. Furthermore, the use of oral amiodarone is considered the standard of care for rhythm management in AF. Prior studies have demonstrated that the administration of a single, oral converting dose of amiodarone has similar rates of sinus rhythm conversion at 24 hours post-intervention compared to Vaughan-Williams Class 1C anti-arrhythmic medications. The use of amiodarone as a first-line therapy for AF is appealing when considering its safety profile.

Objectives: To determine the safety and efficacy of high-dose amiodarone, given as a single uniform oral dose, for the treatment of acute AF in a hospital inpatient setting and acute persistent AF in an outpatient ambulatory clinic.

Methods: This study will be a double-blind randomized controlled trial in patients with symptomatic AF. Amiodarone and placebo capsules will be prepared in single dose packs. A single dose pack will consist of either 2000 mg of amiodarone hydrochloride crushed and placed in 10 gel capsules of 200 mg each, or 10 gel capsules of crushed placebo. Individual dose packs will then be randomly assigned to participants with a unique research number.

Candidate inpatients will be identified through emergency room presentation, outpatient clinic admissions, or inpatient consultation. Once participants have been consented and allocated a study number, they will be randomly assigned a dose pack. Participants will be required to ingest the entire 10 capsule dose pack in one sitting with food witnessed by one of the study investigators or a designated study nurse. Following drug administration, participants will have cardiac monitoring and regular vital sign measurements for up to 48 hours. The investigators will provide the participants with a diary to record any potential adverse side effect symptoms, and the participant will be given the phone number of a study team member to contact if they are concerned about any adverse effects. After the 48 hour period, a study team member will contact the participant and ask specifically about potential adverse events.

Candidate outpatients will be identified through emergency room presentation or outpatient clinics not requiring hospital admission. Once participants have been consented and allocated a study number, they will be assigned a dose pack. Participants will be required to ingest the entire 10 capsule dose pack in one sitting with food. The time of capsule ingestion will be recorded. Following drug administration, participants will be provided with a portable cardiac monitor to wear for 48 hours. History taking of potential adverse side effect symptoms will be performed on a daily basis, or more frequently if required. After the 48 hour period, a 12-lead electrocardiogram with be performed to confirm of successful reversion to sinus rhythm, continuing AF, or other heart rhythm. The portable cardiac monitor will be retrieved and analyzed for evidence of time to successful reversion to sinus rhythm.

The investigators plan to enrol 42 AF patients, with 21 patients randomized to oral amiodarone and 21 patients randomized to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Acute persistent or paroxysmal atrial fibrillation or atrial flutter with duration < 14 days (continuous with no spontaneous conversions), confirmed by ECG or cardiac telemetry
* History of symptoms associated with atrial fibrillation
* Appropriate anticoagulation (warfarin with an international normalized ratio (INR) > 2.0 or direct oral anticoagulant)

Exclusion Criteria:

* Received > 10 g of amiodarone in the prior 6 months, or other Class III anti-arrhythmic agents in the prior 3 months
* previous severe adverse event following a cardioversion for atrial fibrillation
* Hypothyroid and not on thyroid replacement therapy
* Recent myocardial infarction (within 2 weeks)
* Acute pulmonary oedema requiring hospital admission or New York Heart Association (NYHA) class IV heart failure
* Severe left ventricular dysfunction or left ventricular ejection fraction < 36%, as determined by cardiac imaging
* Sick sinus syndrome, high grade atrioventricular block, ventricular rate < 50 beats per minute in the absence of a mechanical pacemaker
* Severe renal or hepatic disease
* Known congenital long QT syndrome
* Hypotension with systolic blood pressure < 90 mmHg
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2026-01-20 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
Time to Successful Reversion to Sinus Rhythm | 48 hours of intervention administration
  Time to successful reversion to sinus rhythm (continuous variable), as documented by continuous cardiac monitoring

SECONDARY OUTCOMES:
Conversion Rate to Sinus Rhythm | 48 hours of intervention administration
  Conversion rate to sinus rhythm (dichotomous variable), as documented by continuous cardiac monitoring
Early Recurrence of Atrial Fibrillation After Initial Reversion to Sinus Rhythm | 48 hours of intervention administration
  Early recurrence of atrial fibrillation (lasting > 6 minutes) after initial reversion to sinus rhythm (dichotomous variable), as documented by continuous cardiac monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD MSCI, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No